CLINICAL TRIAL: NCT02832050
Title: PLAY Therapy Intervention: Re-Modelling Patient Experience (The PLAYTIME Study)
Acronym: PLAYTIME
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: 3 participants screened, all failed screening process
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 197779
Record Dates: First submitted 2016-02-15; First posted 2016-07-13 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Pain; Anxiety; Rheumatology
Keywords: play; therapy
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Play Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The play therapy intervention consists of a standard of care delivered by a play specialist. The play specialist delivers interventions aimed in assisting the child through the process of undergoing procedures. The intervention is semi-structured in order to facilitate a systematic approach which remains individualised and child-centred.
  The intervention requires patients to be classified as 'high risk' or 'low risk' for procedure-related anxiety. This is assessed for all patients at baseline based on parent and clinician opinion. The play specialist may re-classify patients at the initial assessment or at any point whilst working with the child. If this occurs, clear documentation of the rationale for this will be recorded. Patients classified as "high risk" receive additional preparation sessions as detailed in the standard of care.
  Interventions: Behavioral: Play therapy
- Comparator (Placebo Comparator): The comparator group will receive standard care of patients having blood tests within the Trust, which does not include the specific intervention of a play therapist routinely. As part of standard care if a child becomes particularly distressed a clinician may make a decision to refer the child for play therapy. If this occurs during the study period the child will be referred to the play specialist delivering the intervention for the study. The child will then receive play therapy as in the described intervention. They will be excluded from the main analysis but data will still be collected and analysed descriptively.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Play therapy — See previous description of play therapy intervention arm.
  Arms: Intervention
Behavioral: Standard of care — See previous description of comparator arm.
  Arms: Comparator

SUMMARY:
Study synopsis Objectives

* To determine whether delivering a semi-structured play therapy intervention can improve procedure-related anxiety / ability to cope with a procedure / procedure-related pain for children and young people.
* To determine whether delivering a semi-structured play therapy intervention can improve patient experience of blood monitoring.

Patients

* Patients aged 5 - 17 years who are under the care of the rheumatology team.
* Patients expected to require at least two blood tests during a 12 week period. Design
* Recruitment over 24 weeks with each child in the study for a 12 week period.
* 20 patients will receive play therapy intervention as outlined in the play therapy intervention for blood tests.
* 20 patients will be the comparator group. They will be offered standard care for blood tests.
* All children will be offered local anaesthetic cream for each blood test. Blood tests will be performed by venepuncture unless specifically requested otherwise by patient.
* All children will complete outcome measures at baseline, beginning and end of each procedure session and at completion of the study at 16 weeks.

Outcome Measures

* Procedure-related anxiety visual analogue scale (VAS) score - completed by child
* Observer procedure-related anxiety VAS score - completed by parent
* Procedure-related coping VAS score - completed by child
* Procedure-related pain VAS score - completed by child
* Patient experience VAS score - completed by child and parent separately

DETAILED DESCRIPTION:
Children and young people experience significant pain and distress related to procedures. There are many studies looking at psychological and pharmacological interventions demonstrating that these can reduce procedural-related pain and distress. Distraction is frequently studied and consistently demonstrated to reduce procedure-related pain and in some cases distress. It has also been shown that children choose different distractors, and this can be related to age and sex. Best practice for distraction should therefore include identifying and working with individual patient preferences and this can additionally help by giving children some control over the procedure. There are limited studies looking at other interventions such as preparation and parent positioning showing that these interventions can have a positive impact on distress and coping. Few trials examine effect of interventions over time and multiple procedures.

Play specialists provide therapeutic play for children undergoing procedures. They use a combination of psychological interventions alongside pharmacological interventions which includes preparation for the procedure, support during the procedure and post-procedure. However, whilst there is information about what play therapy should involve and which standards should be met, we are unaware of any specific framework of how this should be delivered.

Investigators have developed a semi-structured play therapy intervention, which is developed from standard play therapy theory and well-recognised techniques as well as expert experience. This play therapy intervention is designed to represent a gold standard of care for delivering play therapy to children requiring procedures. The intervention aims to deliver play therapy in a standardised fashion whilst utilising the skill of the play specialist to choose and implement techniques in an individualised approach to each child.

This study aims to deliver this semi-structured play therapy intervention and examine its impact on procedure-related anxiety, coping, pain and patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Child or young person aged 5 to 17 years of age.
* Child under the care of the paediatric rheumatology team at Alder Hey Children's NHS Foundation Trust.
* Child must be expected to require at least 2 blood tests during the study period of 16 weeks as part of their routine care. All decisions regarding requirement for blood tests and/or procedures will be made solely on clinical grounds and not determined in any way by the study team.
* Sufficient time for assessment visit and preparation prior to first procedure.
* The parent or child if aged above 16 years of age has provided written, informed consent to participate in the study.
* The child aged less than 16 years has provided assent appropriate to their age.

Exclusion Criteria:

* Child unable to understand and complete Visual Analogue Scale (VAS) with support.
* Family unwilling to take part in study.
* Patient has previously received regular play therapy.
* Patient receiving psychology input for procedure-related anxiety or anxiety disorder.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Procedure-related anxiety visual analogue scale (VAS) score - completed by child | 1 year
  Procedure-related anxiety visual analogue scale (VAS) score - completed by child

SECONDARY OUTCOMES:
Observer procedure-related anxiety VAS score - completed by parent | 1 year
  Observer procedure-related anxiety VAS score - completed by parent can improve ability to cope with a procedure.
Procedure-related coping VAS score - completed by child | 1 year
  Procedure-related coping VAS score - completed by child
Procedure-related pain VAS score - completed by child | 1 year
  Procedure-related pain VAS score - completed by child
Patient experience VAS score - completed by child and parent separately | 1 year
  Patient experience VAS score - completed by child and parent separately

CONTACTS AND LOCATIONS:
Overall Officials: Michael Beresford, Principal Investigator — Alder Hey Children's NHS Foundation Trust
Locations (1):
- Alder Hey Children's Hospital, Liverpool, Merseyside, United Kingdom